CLINICAL TRIAL: NCT00465777
Title: Reduced in-Hospital Mortality After Improved Management of Patients Hospitalised With Malaria. A Randomised Trial
Brief Title: Improved Management and in-Hospital Mortality
Acronym: MTV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: Statens Serum Institut (Other); World Health Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PED-MTV-2004
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2007-04-25 (Estimated); Status verified 2007-04

CONDITIONS: Mortality; Malaria
Keywords: malaria; mortality; hospital; incentive; personnel; paediatric
MeSH Terms: conditions — Malaria | interventions — Guideline Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Guideline adherence and financial incentive

SUMMARY:
The study intend to evaluate whether the use of standardised malaria case management protocol plus financial incentives added to the availability of free drugs reduce the case-fatality at the paediatric ward.

DETAILED DESCRIPTION:
Mortality at the national paediatric ward in Guinea-Bissau is very high. During a civil war in 1998/1999 the hospital case fatality (CF) decreased by more than 40%, increasing again after the the war. This was attributed to the available free drugs from the humanitarian aid and food incentives to the personnel. Free emergency kits for treatment of severe malaria was introduced, however the CF did not decline. Therefore, the ward was split into two groups of rooms: intervention and control. All the staff of the ward was trained in the use of a standardised guideline for treatment of severe malaria and randomly assigned to one of the groups. All children hospitalised for malaria received the drug emergency kits. The only difference in the intervention group were the small financial incentives and supervision for strict adherence to the guidelines procedures.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization due to malaria
* Non per os

Exclusion Criteria:

* Consent from parent/caretaker declined

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 950
Dates: Start 2004-12; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
In-hospital case-fatality

SECONDARY OUTCOMES:
Cumulative post-discharge mortality on day 28 and length of hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, DMSc, Study Chair — Bandim Health Project
Locations (1):
- Bandim Health Project, Bissau, Bissau Region, Guinea-Bissau

REFERENCES:
- [Derived] Biai S, Rodrigues A, Gomes M, Ribeiro I, Sodemann M, Alves F, Aaby P. Reduced in-hospital mortality after improved management of children under 5 years admitted to hospital with malaria: randomised trial. BMJ. 2007 Oct 27;335(7625):862. doi: 10.1136/bmj.39345.467813.80. Epub 2007 Oct 22. PMID 17954513